CLINICAL TRIAL: NCT05028166
Title: Individual Patient Compassionate Use of Mirdametinib
Status: Available | Type: Expanded Access
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MEK-NF1-701
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Neurofibromatosis Type 1-Associated Plexiform Neurofibromas; Histiocytic Neoplasm; Other MAP-K Pathway Driven Diseases
Keywords: RASopathies; NF1; Neurofibromatosis; Plexiform Neurofibromas; Langerhans
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma, Plexiform | interventions — mirdametinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Mirdametinib (MEK Inhibitor) — Patients will receive oral mirdametinib.

SUMMARY:
This program is being offered on a patient by patient basis and will require company, Institutional Review Board/Independent Ethics Committee, and applicable competent authority approval.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a serious, debilitating or life-threatening medical condition that cannot be treated satisfactorily with an authorized medicinal product or other available standard treatment options, or all other treatment options have been exhausted.
* Patient does not qualify to participate in an ongoing clinical trial.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult